CLINICAL TRIAL: NCT02849288
Title: Bigfoot Biomedical Clinical Research Center (CRC) Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bigfoot Biomedical Inc. (Industry)
Collaborators: Jaeb Center for Health Research (Other); Profil Institute for Clinical Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TST-10025
Record Dates: First submitted 2016-07-20; First posted 2016-07-29 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Use of the Investigational Bigfoot Type 1 Diabetes Management System (T1DMS)
  Interventions: Device: Bigfoot Biomedical Type 1 Diabetes Management System (T1DMS)

INTERVENTIONS:
Device: Bigfoot Biomedical Type 1 Diabetes Management System (T1DMS) — Automated Insulin Delivery System
  Other Names: T1DMS

SUMMARY:
The trial is designed to assess safety and feasibility of the Bigfoot Biomedical Type 1 Diabetes Management System (T1DMS) in up to 50 participants in a closely monitored Clinical Research Center (CRC) environment.

ELIGIBILITY:
Inclusion Criteria:

1. Insulin dependent type 1 diabetes (T1D) for at least one year
2. Age ≥ 7 years of age
3. Weight ≥ 26 kg
4. HbA1c <10%
5. Total BASAL insulin dose (24 hour cumulative total) that is ≥ 5 units and ≤ 72 units per day
6. Insulin regimen stable on either multiple daily insulin injections (MDI) or insulin infusion pump therapy for ≥ 6 months. Regimen must include basal insulin and the use of a rapid acting analog insulin to cover meals (e.g., Novolog, Humalog or Apidra)

   * For participants on MDI, basal insulin must be either once daily Lantus (Glargine) or once daily Levemir (Detemir). The once daily basal insulin dose must be administered in the evening or at bedtime
7. Able to engage in at least 60 minutes of moderate exercise if ≥ 12 years of age (e.g., walking or biking) and if ≥ 7 and < 12 years of age moderate activity (e.g., walking or active play)
8. Willing and able to refrain from use of any medication containing acetaminophen during participation in the study (from the time of consent until study exit)
9. Willing and able to use Humalog insulin during the CRC admission
10. Able to speak and read English

Exclusion Criteria:

1. Females who are sexually active and able to conceive will be excluded if they are not currently using or agree to continue use for the duration of the study an effective method of contraception as determined by investigator
2. Females who are pregnant or intending to become pregnant during participation in the trial

   • Females who are capable of childbearing must have a negative pregnancy test at the time of the screening visit and the pregnancy test must be repeated at enrollment if it was done > 14 days prior
3. Presence of any condition that in the opinion of the investigator impairs the participant's ability to use the system (e.g.,visual impairment that interferes with ability to read the display)
4. Unable or unwilling to use study devices and follow study procedures including the meal and exercise/ activity challenges in the CRC.
5. A current condition that would prevent the use of a study devices, including blood glucose meter (BGM), continuous glucose monitoring (CGM) or insulin pump (CSII)
6. Current participation within the last 60 days in another clinical research study that involves an intervention

   • Participation in research studies involving data collection only is not an exclusion (e.g.,T1D Exchange Registry)
7. Anticoagulant therapy other than aspirin
8. Severe hypoglycemia resulting in seizure OR loss of consciousness within 30 days prior to enrollment
9. Diabetic ketoacidosis (DKA) requiring treatment in a healthcare facility within 30 days prior to enrollment
10. Current use (defined as within the last 3 months) of any medication intended to lower glucose other than insulin (e.g., use of Metformin, Liraglutide, would be exclusions)
11. Current use (defined as within the last 3 months) of any medication that according to the dose, frequency, and route of administration may result in hyperglycemia in the investigator's judgment (e.g., current use of oral steroids)

    • Regular use of inhaled or intranasal steroids is permitted
12. Presence of significant renal disease as evidenced by the presence of any of the following:

    * Current dialysis therapy
    * Serum creatinine of ≥ 2.0 mg/dL within 30 days of enrollment

    For screening purposes, serum creatinine levels will be tested in participants who meet any of the following criteria:
    * A≥10 year history of T1D
    * Are ≥ 45 years of age
13. Presence or history of clinically significant cardiovascular disease (e.g., myocardial infarction, pacemaker, acute coronary syndrome, therapeutic coronary intervention, coronary bypass or stenting procedure, atrial or ventricular fibrillation, treatment for arrhythmia, stable or unstable angina, episode of chest pain of cardiac etiology with associated ECG changes or positive stress test/ cardiac catheterization, congestive heart failure, or cerebrovascular event)
14. ECG findings that indicate participation in the planned exercise/ activity session would be contraindicated as determined by trained personnel at the respective clinical center(s)

    • For screening purposes, ECGs must be completed within 30 days of enrollment in participants who meet any of the following criteria:
    * A ≥ 10 year history of T1D and ≥ 20 years of age
    * Are ≥ 45 years of age
15. History of adrenal insufficiency
16. A diagnosis of gastroparesis or impaired gastric motility that required pharmacological or surgical treatment
17. Celiac Disease (CD) diagnosed < 12 months ago or CD that is currently inadequately treated as determined by the investigator
18. Current alcohol abuse or eating disorder as determined by the investigator
19. Use or abuse of controlled substances without a prescription in the 6 months prior to enrollment
20. History of hemoglobinopathy, sickle cell disease, or blood dyscrasia; blood transfusion within 3 months of enrollment
21. Hematocrit that is above or below the normal reference range of the lab used within 14 days of enrollment
22. Presence or history of any medical or psychiatric condition, or the use of any medication or therapy, that in the opinion of the investigator may be a contraindication to participation in the study
23. Unstable hypertension, thyroid disease, or depression as evidenced by an adjustment in therapy for the condition within the last 2 months, or as determined by investigator

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Evaluate performance of the algorithm/ system commanded delivery of insulin in response to glucose trends from the CGM. in an effort to avoid hypoglycemia and hyperglycemia. | Data will be evaluated upon completion of an individual participant (data collected over approximately 48 hours of use), upon completion of each age cohort, and upon completion of the trial
  Annotated graphs will be used to assess this outcome.
Assessment of safety outcomes and serious adverse events and device related adverse effects. | Data will be evaluated upon completion of an individual participant (data collected over approximately 48 hours of use), upon completion of each age cohort, and upon completion of the trial

SECONDARY OUTCOMES:
Measures of glycemic control | Data will be evaluated upon completion of an individual participant (data collected over approximately 48 hours of use), upon completion of each age cohort, and upon completion of the trial
  Additional measures include but are not limited to, mean glucose (arithmetic and geometric), Glucose variability as assessed by coefficient of variation and standard deviation (arithmetic and geometric). Percentage of time spent below or above glucose threshold levels.
System functionality as evidenced by the availability of CGM data | Data will be evaluated upon completion of an individual participant (data collected over approximately 48 hours of use), upon completion of each age cohort, and upon completion of the trial
  Includes but is not limited to the percentage of time CGM values were available for individual participants and for all participants pooled.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - William Sansum Diabetes Research Institute, Santa Barbara, California
  - Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: Undecided